CLINICAL TRIAL: NCT05772949
Title: Effectiveness of a Smart Hearing Aid on Improving Psychosocial Well-being in Elderly: A Randomized-controlled Trial
Brief Title: Effectiveness of a Smart Hearing Aid on Improving Psychosocial Well-being in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other); Hong Kong Young Women's Christian Association (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: hearing_aid_protocol_v1
Record Dates: First submitted 2023-03-02; First posted 2023-03-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Technology
Keywords: Gerontechnology; Hearing impairment; Hearing aid
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants will be individually randomized to experimental group to use the smart hearing aids from week 1 to week 6, or wait-list control group to follow existing practice (i.e. using no hearing aids or using hearing aids other than the smart hearing aids) from week 1 to week 6 and use the smart hearing aids from week 8 to week 14. A list of random numbers will be generated to create a list of random group allocation (either experimental or wait-list control; allocation ratio 1:1), using the rand function of Excel. The research staff will perform the randomization procedure, by assigning consenting participants who meet all eligibility criteria to the two groups using the list.
Who Masked: Outcomes Assessor
Masking Description: Assessor(s) of the follow-up outcomes and the research analysts will not be involved in the recruitment and intervention delivery and will be blinded to the group allocation (single blindness).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will use the smart hearing aid for 6 weeks.
  Interventions: Device: Experimental group intervention
- Wait-list control group (Experimental): The wait-list control group will follow existing practice (i.e. using no hearing aids or using hearing aids other than the smart hearing aids) for 6 weeks and then use the smart hearing aids for 6 weeks.
  Interventions: Device: Wait-list control group intervention

INTERVENTIONS:
Device: Experimental group intervention — The caregivers will calibrate the smart hearing aids for the participants in the experimental group at the first day of week 1 through the designated mobile application. Caregivers will help the participants to choose the amplification level which best suits their needs.
  Participants in the experimental group can use the smart hearing aids whenever they want during the trial period (i.e. from week 1 to week 6). For participants living in residential setting, caregivers will facilitate them to use the smart hearing aids upon request from the participants or when the caregivers deem the aids beneficial. For participants living in community setting, they will use the smart hearing aids when needed. Their caregivers shall provide assistance in facilitating the participants to use the smart hearing aids. The smart hearing aids do not require any payment from the study participants. They have to return the hearing aids after the study.
  Arms: Experimental group
Device: Wait-list control group intervention — The caregivers will calibrate the smart hearing aids for the participants in the wait-list control group at week 8 through the designated mobile application. Caregivers will help the participants to choose the amplification level which best suits their needs.
  Participants in the wait-list control group will continue the current practice (i.e. using conventional hearing aids or no hearing aids) from week 1 to week 8, and will use the smart hearing aids from week 8 to week 14. Caregivers will facilitate the participants to use the smart hearing aids.
  Arms: Wait-list control group

SUMMARY:
The study has 2 primary research questions, 4 secondary research questions, and 2 auxiliary research questions targeting elderly with hearing impairment. The research questions are:

Primary study questions:

1. Can the use of the smart hearing aids reduce loneliness at the end of intervention?
2. Can the use of the smart hearing aids improve quality of life at the end of intervention?

   Secondary study questions:
3. Can the use of the smart hearing aids improve the communication quality between caregivers and participants at the end of intervention?
4. How is the satisfaction of the participants with the smart hearing aids?
5. What are the factors leading to the use and non-use of the smart hearing aids?
6. What is the usage time of the smart hearing aids?

   Auxiliary study questions:
7. How is the caregiver burden when facilitating the participants to use the smart hearing aids?
8. What are the perceived benefits and acceptability of the smart hearing aids?

DETAILED DESCRIPTION:
Study design

This is a randomised waitlist controlled trial of comparing the outcome indicators between elders using the smart hearing aids for 6 weeks and elders not using the aids. Elders with hearing impairment from District Elderly Community Service, Haven of Hope Christian Service (HOH DECS) and Day Care Centre for the Elderly, Haven of Hope Christian Service (HOH DE) per the verbal or written medical recommendation by doctor, nurse, physiotherapist, occupational therapist or speech therapist, or currently using hearing aids other than the smart hearing aids in the current study. We will also explore the perceived benefits and acceptability of the smart hearing aids of the participants and caregivers.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP) and Declaration of Helsinki.

Subjects

Elders with hearing impairment per the verbal or written medical recommendation by doctor, nurse, physiotherapist, occupational therapist or speech therapist, or currently using hearing aids other than the smart hearing aids in the current study from HOH DECS and HOH DE will be recruited for the main analysis.

Procedures

Caregiver training

Identical training sessions will be delivered to caregivers on calibrating and facilitating the participants to use the smart hearing aids.

Participants' recruitment and consent

In the study sites, the staff will invite eligible residents and members to join the trial. Residents scoring above the cutoff for dementia in Montreal Cognitive Assessment (MoCA) and not receiving a medical diagnosis of dementia or other mentally incapacitating disease will be classified as competent in giving consent. For elders scoring below the cutoff in MoCA or receiving a diagnosis of mentally incapacitating disease, we will follow the criteria stated in the Alzheimer Europe Report (2011) to ensure that they are provided chances to give consent. In particular, four criteria will be evaluated, including 1) the person must have sufficient capacity to understand the information, 2) the person is able to retain, use and weight up such information for making a decision, 3) the person will understand the benefit, risk, and convenience, 4) the person must have the ability to communicate the decision. The University of Hong Kong (HKU) research staff and the care staff will first commit them in a causal chat to assess their ability to communicate and understand the dialogues.

If residents / members are competent in giving consent, both residents / members and their family members will be approached for consent. In cases residents are not competent in giving consents, only their family members will be approached for consent. They will then be referred to join a 1-to-1 study introduction session. In this session, HKU research staff and service unit staff will introduce the study to the participant, and invite them to sign a consent form. As a voluntary participation, the participants have the right to withdraw from the study and intervention any time without consequences.

For caregivers, written informed consent will be obtained before doing qualitative interview.

Baseline assessment

After the consent is obtained, the HKU research staff will assist the participants to complete UCLA Loneliness Scale 3-item (UCLA 3-item), World Health Organization Quality of Life Brief Version (WHOQOL-BREF), and Satisfaction with Amplification in Daily Life (SADL) (if they currently use other brands of hearing aids).

Randomization

Participants will be individually randomized to experimental group to use the smart hearing aids from week 1 to week 6, or wait-list control group to follow existing practice (i.e. using no hearing aids or using hearing aids other than the smart hearing aids) from week 1 to week 6 and use the smart hearing aids from week 8 to week 14. A list of random numbers will be generated to create a list of random group allocation (either experimental or wait-list control; allocation ratio 1:1), using the rand function of Excel. The research staff will perform the randomization procedure, by assigning consenting participants who meet all eligibility criteria to the two groups using the list.

Calibration

The caregivers will calibrate the smart hearing aids for the participants in the experimental group at the first day of week 1 and the wait-list control group at week 8 through the designated mobile application. Caregivers will help the participants to choose the amplification level which best suits their needs.

Implementation

Participants in the experimental group can use the smart hearing aids whenever they want during the trial period (i.e. from week 1 to week 6). For participants living in residential setting, caregivers will facilitate them to use the smart hearing aids upon request from the participants or when the caregivers deem the aids beneficial. For participants living in community setting, they will use the smart hearing aids when needed. Their caregivers shall provide assistance in facilitating the participants to use the smart hearing aids. The smart hearing aids do not require any payment from the study participants. They have to return the hearing aids after the study.

Participants in the wait-list control group will continue the current practice (i.e. using conventional hearing aids or no hearing aids) from week 1 to week 8, and will use the smart hearing aids from week 8 to week 14. Caregivers will facilitate the participants to use the smart hearing aids.

Data collection

HKU research staff who is blinded to the group allocation will administer all the questionnaire in assessing the primary outcomes. For the experimental group, the questionnaire assessing the primary outcomes and the secondary outcomes of communication quality and satisfaction with the hearing aids will be administered at baseline and week 6. HKU research staff will conduct questionnaire exploring the secondary outcomes of factors leading to the use and non-use of the smart hearing aids, usage time with caregivers and participants and the auxiliary outcome of caregiver burden at week 1, week 3, and week 6. For wait-list control group, the questionnaire assessing the primary outcomes will be administered at baseline, week 6 and week 14. The questionnaire exploring the secondary and auxiliary outcomes will be conducted by HKU research staff with caregivers and participants at week 8, week 10, and week 14.

In case of events (e.g. COVID-19) that prohibit HKU research staff from conducting assessment on site, assessment will be conducted via online communication apps (e.g. Zoom).

Qualitative interview

To collect feedback towards the smart hearing aids, we will use purposive sampling to select 10 - 15 participants and 4 - 8 caregivers to conduct semi-structured qualitative interviews to collect opinion on their perceived acceptance and benefits on the features of the smart hearing aids. An interview guide with open-ended and iterative questions will be used to probe for more experiences from the interviewees. Each interview will be conducted by a trained research assistant and will last about 30 minutes.

Blinding

Participants and caregivers cannot and will not be blinded to the intervention. Assessor(s) of the follow-up outcomes and the research analysts will not be involved in the recruitment and intervention delivery and will be blinded to the group allocation (single blindness).

Sample size determination

The sample size is estimated by the current number of elders with hearing impairment and / or currently using hearing aids other than the smart hearing aids used in this study in the test sites. In the HOH DECS, 10 elders have been diagnosed hearing impairment and / or are using hearing aids other than the smart hearing aids used in the study. In the HOH DE, 20 have been diagnosed or are using other hearing aids. Therefore, the study will include 30 elders in total.

With reference to Nieman et al. (2022), the between group change difference on UCLA loneliness scale (20-item version) is 2.26 with a pooled variance of 61.9. Using the sample size calculation formula in Noordzij et al. (2010), Type 1 error rate of 5% and power 80%, the number of participant required for each group, 18 participants are required in each group for analysis. Assuming attrition rate of 5%, at least 20 participants need to be recruited.

Data analyses

Main analysis

Linear mixed model analysis will be used to test the interaction between group and time. A partial-eta square will be used to estimate the effect size of the outcome indicators in comparing the intervention group with the wait-list control group. Dependent sample t-test will be used to investigate the within group effects based on the data from both experimental and wait-list control group.

Process evaluations

For the quantitative secondary outcomes, descriptive statistics will be used to show the opinions. For the qualitative secondary outcomes, the content will be analyzed using framework analysis to construct a coherent and logical structure from the classification of many opinions.

Qualitative interview

The interview content will be transcribed verbatim in Chinese for further analysis. We will analyze the qualitative interview transcripts using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions on the use of the smart hearing aids. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for participants:

* With hearing impairment per the verbal or written medical recommendation by doctor, nurse, physiotherapist, occupational therapist or speech therapist, or currently using hearing aids other than the smart hearing aids in the current study, and
* Able to understand Chinese

Inclusion criteria for caregivers:

* Responsible for helping the participants to use the smart hearing aids, and
* Able to understand Chinese

Exclusion Criteria:

Exclusion criteria for participants:

* Unable to use the hearing aids independently, and
* Unable to use the hearing aids with caregivers' assistance, or
* Ménière's disease, or
* Deafness (i.e. cannot hear speech, even when the speaker is talking loudly next to the better hearing ear)

Exclusion criteria for caregivers:

• Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
6-week change in loneliness after using the smart hearing aids for 6 weeks | Baseline, the 6th week and the 14th week (waitlist control group only)
  Change of loneliness after using the smart hearing aids for 6 weeks will be measured by UCLA Loneliness Scale 3 items (UCLA 3-items, Russell et al., 1980; Liu et al., 2020). The minimum and maximum values of the scale are 3 and 9 respectively, with higher score indicating higher level of loneliness.
6-week change in quality of life after using the smart hearing aids for 6 weeks | Baseline, the 6th week and the 14th week (waitlist control group only)
  Change in quality of life after using the smart hearing aids for 6 weeks will be measured by World Health Organization Quality of Life Brief Version (WHOQOL-BREF, World Health Organization, 2004).The minimum and maximum values of the scale are 26 and 130 respectively, with higher score indicating poorer quality of life.

SECONDARY OUTCOMES:
6-week change in communication quality between participants and caregivers | The 1st week, the 3rd week and the 6th week of using the smart hearing aids
  Caregivers will complete eight items indicating the communication quality with participants to use the smart hearing aids on a 5-point Likert scale (i.e. 1 indicating strongly disagree and 5 indicating strongly agree) in the past week at week 1, 3 and 6. The minimum and maximum values of the scale are 8 and 40 respectively, with higher score indicating higher level of communication quality.
6-week change in the elders' satisfaction after using the smart hearing aids for 6 weeks | Baseline, the 6th week and the 14th week (waitlist control group only)
  Change of elders' satisfaction after using the smart hearing aids for 6 weeks measured by Satisfaction with Amplification in Daily Life (SADL, Cox & Alexander, 1999; Veiga et al., 2005; Kam, 2012). The minimum and maximum values of the scale are 12 and 84 respectively, with higher score indicating higher level of satisfaction.
Qualitative Measure: Factors leading to the use and non-use of the smart hearing aids during the 6-week trial period | The 1st week, the 3rd week and the 6th week of using the smart hearing aids
  Participants or caregivers will complete three items indicating the factors leading to the use and non-use of the smart hearing aids in the past week at week 1, 3 and 6.
The usage time of the smart hearing aids during the 6-week trial period | The 1st week, the 3rd week and the 6th week of the trial period
  Participants or caregivers will report the average usage time of the smart hearing aids in the past week at week 1, 3 and 6
6-week change in caregivers burden while facilitating the use of the smart hearing aids | The 1st week, the 3rd week and the 6th week of the trial period
  Caregivers will complete an item indicating their burden in facilitating the participants to use the smart hearing aids on a 5-point Likert scale (i.e. 1 indicating no burden and 5 indicating severe burden) at week 1, 3 and 6.
Qualitative Measure: Perceived benefits and acceptability of the smart hearing aids of participants | Within 2 weeks after the participants using the smart hearing aids for 6 weeks
  The participants answer the following questions in semi-structured qualitative interviews:
  1. Do you like the appearance of the smart hearing aids?
  2. Is the smart hearing aids easy to use?
  3. Is it comfortable to wear the smart hearing aids?
  4. Are you satisfied with the sound amplification of the smart hearing aids?
  5. Do you think the use of the smart hearing aids help you communicate with others?
  6. Do you like the smart hearing aids?
  7. Do you want to continue to use the smart hearing aids in the future?
Qualitative Measure: Perceived benefits and acceptability of the smart hearing aids of caregivers. | Within 2 weeks after the participants using the smart hearing aids for 6 weeks
  The caregivers answer the following questions in semi-structured qualitative interviews:
  1. Compared to traditional hearing aids, do you think the appearance of the smart hearing aids (hereafter refers as the aids) could appeal the elders to wear it?
  2. How is the size of the aids?
  3. Is it easy to use the aids?
  4. To what extent, did you expect the elders would use the aids?
  5. To what extent, are the elders willing to use the aids?
  6. Did the use of the aids improve the communication quality between the elders and you?
  7. Did the elders become more proactive to socialize with others after the use of the aids?
  8. Did you discover other benefits due to the use of the aids?
  9. What were your concerns when you were asked to help the elders to use the aids?
  10. Did you discover these concerns when helping the elders to use the aids?
  11. On the whole, are you satisfied with the aids?
  12. To what extent, do you want the elders to continue to use the aids?

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, Principal Investigator — The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Haven of Hope Day Care Centre for the Elderly, Hong Kong
  - Haven of Hope District Elderly Community Service, Hong Kong
  - Hong Kong Young Women's Christian Association Wan Wah Care and Attention Home for the Elderly, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Background] Cox RM, Alexander GC. Measuring Satisfaction with Amplification in Daily Life: the SADL scale. Ear Hear. 1999 Aug;20(4):306-20. doi: 10.1097/00003446-199908000-00004. PMID 10466567
- [Background] Kam AC. Hearing-aid outcomes in Chinese adults: clinical application and psychometric properties of the Chinese version of the Satisfaction with Amplification in Daily Life questionnaire. Int J Audiol. 2012 Jun;51(6):450-5. doi: 10.3109/14992027.2012.670732. Epub 2012 Apr 26. PMID 22537034
- [Background] Liu T, Lu S, Leung DKY, Sze LCY, Kwok WW, Tang JYM, Luo H, Lum TYS, Wong GHY. Adapting the UCLA 3-item loneliness scale for community-based depressive symptoms screening interview among older Chinese: a cross-sectional study. BMJ Open. 2020 Dec 10;10(12):e041921. doi: 10.1136/bmjopen-2020-041921. PMID 33303463
- [Background] Nieman CL, Betz J, Garcia Morales EE, Suen JJ, Trumbo J, Marrone N, Han HR, Szanton SL, Lin FR. Effect of a Community Health Worker-Delivered Personal Sound Amplification Device on Self-Perceived Communication Function in Older Adults With Hearing Loss: A Randomized Clinical Trial. JAMA. 2022 Dec 20;328(23):2324-2333. doi: 10.1001/jama.2022.21820. PMID 36538311
- [Background] Noordzij M, Tripepi G, Dekker FW, Zoccali C, Tanck MW, Jager KJ. Sample size calculations: basic principles and common pitfalls. Nephrol Dial Transplant. 2010 May;25(5):1388-93. doi: 10.1093/ndt/gfp732. Epub 2010 Jan 12. PMID 20067907
- [Background] Piau A, Campo E, Rumeau P, Vellas B, Nourhashemi F. Aging society and gerontechnology: a solution for an independent living? J Nutr Health Aging. 2014 Jan;18(1):97-112. doi: 10.1007/s12603-013-0356-5. PMID 24402399
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Veiga LR, Merlo AR, Mengue SS. Satisfaction level with hearing aid in the daily life of Army Healthcare System users. Braz J Otorhinolaryngol. 2005 Jan-Feb;71(1):67-73. doi: 10.1016/s1808-8694(15)31287-8. Epub 2006 Jan 2. PMID 16446894